CLINICAL TRIAL: NCT01328132
Title: Effect of Hyperoncotic Albumin on Vascular Hemodynamics and Oxygen Delivery Following Orthotopic Liver Transplant
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Sheldon Magder, MD, McGill University Health Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10-287-BMA
Record Dates: First submitted 2011-03-31; First posted 2011-04-04 (Estimated); Last update posted 2011-04-04 (Estimated); Status verified 2011-01

CONDITIONS: Other Complications of Liver Transplant
Keywords: Liver; transplant; albumin
MeSH Terms: interventions — Sodium Chloride; Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saline (Active Comparator)
  Interventions: Drug: Saline
- 25% albumin (Experimental)
  Interventions: Drug: 25% albumin

INTERVENTIONS:
Drug: Saline — 100 ml of saline will be given in addition to the standard of care every 8 hours for 24 hours.
  Arms: Saline
Drug: 25% albumin — 100 ml of 25% albumin will be given in addition to the standard of care every 8 hours for 24 hours
  Arms: 25% albumin

SUMMARY:
The primary aim of this study is to assess the effect of hyperoncotic albumin on vascular hemodynamics and oxygen delivery after orthotopic liver transplant. The secondary aim is to try to identify the dominant physiological mechanism so that we will be able to better identify patients that may benefit from the use of albumin (25%) boluses in addition to standard care in patients following liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Patients from the Critical care Unit
* Patients with a pulmonary artery occlusion catheter Inclusion:patients immediately following liver transplantation

Exclusion Criteria:

* Patients not giving informed consent
* Patients who have received > 300 ml of albumin within 24 hours prior to inclusion
* Patients known to have previous adverse reaction to human albumin solution
* Patients who have religious restriction to receive human blood products
* Patient who have initial graft failure
* Patients with fluctuating hemodynamics
* Concerns of the treating surgeon

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Cardiac index (CI) | 60 minutes after the infusion of the fluid

SECONDARY OUTCOMES:
Cardiac function response | 30 and 60 minutes after the infusion of the fluid
  An improvement in Q due primarily to a change in cardiac function should have an increase in Q of ≥ 0.3 ml/min/m2/mmHg
A decrease in leak and plasma expansion | 30 and 60 minutes after the infusion of the fluid
  A decrease in leak and plasma expansion will be determined by the Harrison formula for calculating a change in plasma volume from the change in Hb and change in Hct
Cardiac output response | 30 and 60 minutes after the infusion of the fluid
  Cardiac output response primarily due to a "volume effect" would be expected to have an increase of CVP of a minimum of 2 mmHg and an increase in CI of > 0.3 L/min/m2 per mmHg.
Detoxification effect of albumin | 30 and 60 minutes after infusion
  A increase in vascular tone will be identified by an increase in systemic vascular resistance or a rise in blood pressure without a change in cardiac output or a rise in blood pressure with a fall in cardiac output

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Magder, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Royal Victoria Hospital, Montreal, Quebec, Canada